CLINICAL TRIAL: NCT06195189
Title: Sunvozertinib Combined With Chemotherapy for EGFRm + Locally Advanced or Metastasis NSCLC Patients After EGFR-TKI Treatment Failure：Phase I/II (WU-KONG36)
Brief Title: Sunvozertinib Combined With Chemotherapy for EGFRm After EGFR-TKI Treatment Failure：Phase I/II
Acronym: WU-KONG36
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Oncology, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2023EI002
Record Dates: First submitted 2023-12-24; First posted 2024-01-08 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Sunvozertinib; EGFR; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunvozertinib combined with chemotherapy (Pemetrexed +platinum) (Experimental): Sunvozertinib 200mg Quaquedie (QD) combined with chemotherapy (Pemetrexed +platinum)
  Interventions: Drug: Sunvozertinib; Drug: Chemotherapy

INTERVENTIONS:
Drug: Sunvozertinib — Sunvozertinib 200mg Quaquedie (QD)
Drug: Chemotherapy — Pemetrexed +platinum

SUMMARY:
To access the anti-tumor efficacy, safety and tolerability of Sunvozertinib combined with chemotherapy in patients with locally advanced or metastatic non-small-cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) sensitizing mutations who have progressed following standard TKI therapy.

DETAILED DESCRIPTION:
This study is a single arm study to access the anti-tumor efficacy, safety and tolerability of Sunvozertinib combined with chemotherapy in patients with locally advanced or metastatic non-small-cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) sensitizing mutations who have progressed following standard TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

1. To provide a signed and dated, written informed consent.
2. 80≥Age ≥ 18 years old
3. Histologically or cytologically confirmed non-squamous NSCLC with documented EGFR mutations from a local laboratory
4. EGFR-sensitive mutations including exon 19 deletion and exon 21 L858R mutated, and exon 20 T790M mutated.
5. Predicted life expectancy ≥ 12 weeks
6. EGFR-TKI resistance or intolerant to standard EGFR TKIs therapy.
7. No previous systemic chemotherapy for advanced or metastatic disease.
8. Adequate organ system function:
9. Patient must have measurable disease according to RECIST 1.1.
10. Patients with stable or pre-treated brain metastasis (BM) can be enrolled

Exclusion Criteria:

1. Spinal cord compression or meningeal metastasis
2. A history of malignant tumors within 2 years.
3. With known resistant mutations that have approved target therapy
4. Recover from AEs caused by previous treatment
5. A history of stroke or intracranial hemorrhage within 6 months prior to initial dosing.
6. Any severe or poorly controlled systemic disease per investigator's judgment active infections, including but not limited to hepatitis B (HBV), hepatitis C (HCV), and human immunodeficiency (HIV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Time from first dose to last dose, or up to 24 month
  To assess sunvozertinib overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)

SECONDARY OUTCOMES:
Duration of Response (DoR) | Time from first subject dose to study completion, or up to 36 month
  To assess duration of response for subjects with CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator , defined as the time from the first documented CR or PR to disease progression or death
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month
  To assess progression-free survival of patients treated by sunvozertinib according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as first dose to first documented disease progression assessed by investigator or death due to any cause
Overall survival (OS) | Time from first subject dose to study completion, or up to 36 month
  To assess overall survival, define as first dose to the death of the subject due to any cause
Adverse events (AEs) according to CTCAE 5.0 | From first dose until 28 days after the last dose, up to 24 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No